CLINICAL TRIAL: NCT03200080
Title: A Randomized, Double-Blind, 6-Way Crossover Study to Determine the Abuse Potential of Tozadenant Relative to D-Amphetamine and Placebo When Administered Orally in Healthy, Non-Dependent, Recreational Polydrug Users With Stimulant Experience, Under Fed Conditions
Brief Title: A Study to Determine the Abuse Potential of Tozadenant Relative to D-Amphetamine and Placebo When Administered Orally in Healthy, Non-Dependent, Recreational Polydrug Users
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New Safety Information
Sponsor: Biotie Therapies Inc. (Industry)
Collaborators: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: TOZ-CL09
Record Dates: First submitted 2017-03-14; First posted 2017-06-27 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2017-06

CONDITIONS: Abuse Potential
MeSH Terms: interventions — tozadenant; Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment A (Placebo Comparator): Placebo oral tablet and Placebo oral capsule
  Interventions: Drug: Placebo oral tablet; Drug: Placebo oral capsule
- Treatment B (Experimental): Tozadenant 120 mg
  Interventions: Drug: Tozadenant; Drug: Placebo oral capsule
- Treatment C (Experimental): Tozadenant 240 mg
  Interventions: Drug: Tozadenant; Drug: Placebo oral capsule
- Treatment D (Experimental): Tozadenant 480 mg
  Interventions: Drug: Tozadenant; Drug: Placebo oral capsule
- Treatment E (Active Comparator): d-amphetamine 20 mg
  Interventions: Drug: Placebo oral tablet; Drug: d-amphetamine
- Treatment F (Active Comparator): d-amphetamine 40 mg
  Interventions: Drug: Placebo oral tablet; Drug: d-amphetamine

INTERVENTIONS:
Drug: Tozadenant — 2, 4, 6 or 8 Tozadenant 60 mg tablets
  Other Names: SYN115
  Arms: Treatment B; Treatment C; Treatment D
Drug: Placebo oral tablet — 2, 4, 6 or 8 Tozadenant matching placebo tablets
  Arms: Treatment A; Treatment E; Treatment F
Drug: d-amphetamine — 2 or 4 capsules, each containing 2 over-encapsulated d-amphetamine 5 mg tablets
  Arms: Treatment E; Treatment F
Drug: Placebo oral capsule — 2 or 4 capsules, each containing d-amphetamine matching over-encapsulated PLACEBO 200 mg lactose tablet
  Arms: Treatment A; Treatment B; Treatment C; Treatment D

SUMMARY:
This will be a single-dose, randomized, double-blind, active- and placebo-controlled, double dummy, 6-way crossover study to determine the abuse potential of tozadenant relative to d-amphetamine and placebo, when administered orally in healthy non-dependent, recreational polydrug users with stimulant experience, under fed conditions.

Each subject will participate in a medical Screening visit, a 4-day (3-night) qualification (drug discrimination) visit, six 3-day (2-night) treatment periods, and a follow-up visit.

DETAILED DESCRIPTION:
The Qualification Phase will be conducted as a single, 4-day visit. Doses will be administered in a randomized, double-blind crossover manner following administration of a standard low-fat meal. Subjects will be dosed with 20 mg of d-amphetamine or matching placebo d-amphetamine on Day 1 and Day 2, approximately 24 hours apart. PD assessments will be conducted before dosing and at time points for up to 8 hours post dosing. Safety assessments will be conducted before dosing and for at least 24 hours following dosing. Data will be reviewed to determine subject eligibility.

The last drug administration in the Qualification Phase and the first drug administration in the Treatment Phase will be separated by a washout interval of at least 7 days and not to exceed 28 days.

During the Treatment Phase, there will be 6 treatment periods; subjects will receive a single oral dose of each of the following treatments with applicable matching oral placebos in a randomized, double-blind, double-dummy fashion following the administration of a standard, low-fat meal. The following treatments will be administered:

* Treatment A: placebo (matched to tozadenant and d-amphetamine)
* Treatment B: tozadenant 120 mg
* Treatment C: tozadenant 240 mg
* Treatment D: tozadenant 480 mg
* Treatment E: d-amphetamine 20 mg
* Treatment F: d-amphetamine 40 mg

Drug administration will occur on Day 1 of each of the 6 treatment periods. PD and PK assessments will be collected during the 24 hours post-dose and safety assessments will be collected during the 36 hours post-dose. Subjects will be discharged on Day 2, after approximately 36 hours post-dose, or remain at the clinical research unit longer (e.g., 48 hours or until the following morning) if there are safety concerns, at the discretion of the investigator or designee. Drug administration in each treatment period will be separated by a washout interval of at least 7 days after the last dose of study drug.

Subjects will return for an end-of-study safety Follow-up visit approximately 7 to 14 days after the subject's last study drug dose in the Treatment Phase or following early withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects 18 to 55 years of age, inclusive.
* Have a body mass index (BMI) within the range of 18.0 to 30.0 kg/m2 and a minimum weight of at least 50.0 kg
* Current recreational polydrug users who self-report to:

  * Have used stimulants (e.g., amphetamines, cocaine, methylphenidate) for non-therapeutic purposes (i.e., for psychoactive effects) at least 10 times in the past year and at least 1 time in the 8 weeks before Screening.
  * Have at least 10 lifetime uses of drugs (e.g., opioids, sedatives) from at least 1 other class other than alcohol.
* Agree to use an approved method of contraception
* Be willing and able to abide by all study requirements and restrictions
* Additional criteria may apply

Exclusion Criteria:

* Substance or alcohol dependence within the past 2 years,
* Clinically significant medical history or illness
* Female subjects who have a positive pregnancy test, are currently pregnant or lactating, or who are planning to become pregnant within 30 days of last study drug administration.
* Donation or loss of more than 500 mL whole blood within 30 days preceding the Screening visit.
* Additional criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Drug Liking | 24 hours
  Drug Liking Visual Analog Scale (VAS) ("at this moment"), assessed on a bipolar, 0- to 100-point visual analog scale.

SECONDARY OUTCOMES:
Balance of effects | 24 hours
  Based on Drug Liking VAS
Global effects | 24 hours
  Overall Drug Liking VAS
Positive drug effects | 24 hours
  High VAS
Positive drug effects | 24 hours
  Good Drug Effects VAS
Negative drug effects | 24 hours
  Bad Drug Effects VAS
Stimulant effects | 24 hours
  Alertness/Drowsiness VAS
Stimulant effects | 24 hours
  Agitation/Relaxation VAS
Other drug effects: | 24 hours
  Hallucinations VAS
Other drug effects: | 24 hours
  Detached VAS
Other drug effects: | 24 hours
  Addiction Research Center Inventory (ARCI)
Other drug effects: | 12 hours
  Drug Similarity VAS
Other drug effects: | 24 hours
  Bowdle VAS
Cognitive and psychomotor effects | 24 hours
  Divided Attention Test
Cognitive and psychomotor effects | 24 hours
  Choice Reaction Time

CONTACTS AND LOCATIONS:
Overall Officials: Michael McDonnell, MD, Principal Investigator — INC Research Toronto
Locations (1):
- INC Research Toronto, Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No